CLINICAL TRIAL: NCT06887543
Title: The Impact of Time Restricted Eating on Type 2 Diabetes Study
Brief Title: The Impact of Time Restricted Eating on Type 2 Diabetes
Acronym: EaT2DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: clinical facility could no longer support study conduct; loss of funding, PI left the institution
Sponsor: Rockefeller University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Jose O. Aleman, MD PhD, Principle Investigator, Rockefeller University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: JAL-1056
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Time restricted eating; Intermittent fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted eating (Active Comparator): Selection of the order of the arms is randomized prior to active study participation. Caloric requirements and meal selection are done during screening and calculated to maintain weight neutrality. In Arm 1, participants are required to start breakfast at 8 AM, complete lunch by 2 PM (80% of total daily calories) and snack by 4 PM (20% of calories). They then fast from 4 PM till 8 AM the next day (16 hour fast). This is done for six days. The next day is for testing (2 hour oral glucose tolerance test, resting energy expenditure, research and clinical blood tests) prior to crossover to Arm 2.
  Interventions: Other: Meal timing; Other: Time restricted eating
- Usual feeding pattern, with meals eaten ad lib (Placebo Comparator): Participants consume the same meals as in the other arm, but may eat ad lib without prolonged fasting. This is done for six days. Post-testing including 2 hour oral glucose tolerance test, resting energy expenditure, and research and clinical blood tests are done the following day.
  Interventions: Other: Usual feeding pattern.

INTERVENTIONS:
Other: Meal timing — Participants either eat all of their daily calories between 8 AM and 4 PM with 16 hours fasting for six days, or they eat the same meals ad lib daily for six days. After post-testing, they crossover to the other arm.
  Arms: Time restricted eating
Other: Time restricted eating — Eating restricted to 8 AM - 2 PM for 80% of caloric intake, the remaining 20% consumed by 4 PM, subsequent 16-hour fasting (4 PM-8 AM) each day for six days while on Time Restricted Arm.
  Arms: Time restricted eating
Other: Usual feeding pattern. — Participant consumes usual diet ad lib without enforced fasting period for six days while on Usual Feeding Pattern arm.
  Arms: Usual feeding pattern, with meals eaten ad lib

SUMMARY:
Time-restricted feeding limits caloric intake to active daytime hours with fasting for 14 to 16 hours. It has shown great promise as a novel intervention for stabilizing blood glucose, reducing weight, and improving cardiovascular disease outcomes. However, this approach has not been tested on people with diabetes, a group that would benefit from improved blood glucose and weight loss.

The impact of Time-Restricted Eating on Type 2 Diabetes Study (EaT2D Study) is a randomized six-day weight stable crossover feeding study in the Day Patient/Outpatient unit of The Rockefeller Hospital investigating how the time of day that meals are eaten affects weight, blood sugar and blood pressure. The investigators will compare an early time-restricted eating intervention (80% of calories consumed before 2 pm) to a usual feeding pattern (50% of calories consumed after 4 pm) among 10 persons with type 2 diabetes to determine effects on blood sugar and small molecules found in the blood.

Studies have shown benefits of eating during active periods (mornings and early afternoon) for metabolic health (blood sugar, body weight) compared to eating during inactive periods (evening and bedtime). Eating earlier in the day may lead to reduced sugar stores, burning fat for energy, and decreased inflammation when compared to eating later in the day. The investigators will compare the effects of eating earlier during the day for six days versus later in the day for six days, on blood sugar, blood pressure, blood ketones, and other measures of metabolic health in diabetic participants. Studies in animals supports these benefits.

DETAILED DESCRIPTION:
Early Time Restricted Eating (eTRE) is a meal timing strategy that restricts the daily eating window to the first 6-8 waking hours of the day, while extending the fasting window between the final meal of the day and the first meal the following morning.

There is an increasing body of evidence that circadian misalignment caused by changes in sleeping and eating behaviors is a significant contributor to obesity and cardiometabolic disease, and late-night eating behaviors are associated with obesity, weight loss inhibition, and various cardiovascular disease risk factors. While the mechanisms underlying these correlations are not well understood, these effects are most likely due to suboptimal timing of caloric intake against diurnal variations in hormone and metabolite activity. Therefore, eTRE shows great promise as a novel intervention for addressing obesity and related cardiovascular outcomes. In support of this, recent studies have demonstrated weight-independent benefits of eTRE on measures of insulin sensitivity and cardiac risk. However, studies to date have primarily focused on metabolically healthy or prediabetic populations and the effect of this dietary practice on individuals with type 2 diabetes has not yet been evaluated.

To this end, the investigators propose to conduct a randomized isocaloric 15-day crossover feeding trial in the outpatient unit at The Rockefeller University Hospital (RUH) comparing an eTRE intervention (feeding window 8 AM-4 PM; 80% of calories consumed prior to 2 PM; remaining 20% to be consumed by 4 PM) to a Usual Feeding Pattern (UFP) (50% of calories consumed after 4 PM) among 10 persons with type 2 diabetes and obesity to determine effects on glycemic variation and various time-in-range metrics. The primary hypothesis of this study is that restriction of caloric intake to earlier in the day will have metabolic benefits in terms of glycemic variation and time in hyperglycemia relative to consuming the majority of calories later in the day, as in the control arm. Additionally, the investigators anticipate no increase in hypoglycemia in the eTRE arm compared to the UPF control arm. This feeding study provides a unique opportunity to study the weight-independent effects of eTRE on a population that has frequently been excluded from dietary studies in this area, yet for whom diet and lifestyle modifications are foundational components of treatment. Additionally, the proposed work will complement our recent study performed at Rockefeller University Hospital (RUH), "The Time-Restricted-Feeding Effects on Inflammation and Obesity" (TRIO) Study, which utilized a similar study design to show the weight-independent glycemic benefits of eTRE in individuals with prediabetes and obesity.

The investigators propose to obtain glucometric data including glycemic variation and various time in range metrics by Continuous Glucose Monitoring (CGM), circulating advanced glycation end-products (AGEs), and targeted plasma metabolomic profiles as surrogate measures of overall dysglycemia affected by the eTRE intervention in the RUH metabolic study.

The collaborative research proposed between RUH and New York University (NYU) Obesity Center in this application will take advantage of the expertise of both centers and advance the science of obesity and cardiovascular disease. Members of our team have extensive experience in clinical dietary studies and advanced glucometric analysis. The investigators will be able to evaluate the effectiveness of eTRE as a weight-independent therapeutic strategy for type 2 diabetes management and identify the metabolic pathways invoked, thereby synergistically expanding the work of each institution.

The rationale for this study is that early time-restricted eating (eTRE) has been shown to improve glycemic variation in a weight-neutral setting within 48 hours in individuals with prediabetes, making it a promising dietary intervention to mitigate dysglycemia. However, it has not been studied in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 able to give consent
2. BMI >25 kg/m2
3. Hemoglobin A1C ≥ 6.5%
4. Willing to eat only the food provided
5. Willing to follow the feeding schedule, including fasting for 16 hours/day for six days.
6. Usual sleep time is between 10 PM and 8 AM
7. Fluent in the English language

Exclusion Criteria:

1. Current use of anti-obesity medications (Ozempic, Mounjaro, Trulicity, Wegovy, Zepbound, Qsymia, Contrave, Saxenda, Victoza, Orlistat)
2. Report history of Cirrhosis
3. HIV positive
4. Self-reported autoimmune disease (rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease, ulcerative colitis, psoriasis, etc.)
5. Current use of steroids (inhalers are permissible)
6. Currently pregnant
7. Smoked tobacco within the last 3 months
8. Allergy to adhesive tape
9. Skips breakfast
10. Followed TRF or intermittent fasting in the last 2 weeks
11. Shift or night worker
12. Current use of insulin
13. Current use of sulfonylureas
14. Current use of glucagon-like peptide-1 (GLP-1) receptor agonists
15. Hemoglobin A1c >8%
16. Unable to sync smartphone with Bluetooth for scale data
17. Any medical, psychological, or social condition that, in the opinion of the investigator, would jeopardize the health or well-being of the participant during any study procedures or the integrity of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Change in glycemic variation by Mean Amplitude of Glycemic Excursion (MAGE) in the Early Time Restricted Eating (eTRE) arm relative to the usual feeding pattern (UFP) arm between Day 1, Day 8, and Day 15. arm | From Day 1-15 of study intervention.
  Glycemic variation (changes in glucose levels in milligrams per deciliter (mg/dL) will be measured by continuous glucose monitoring (Abbott Freestyle Libre) recorded every 5 minutes for the entire study, as well as 2-hour oral glucose tolerance testing (measured by glucose measurements in mg/dL every 30 minutes for 120 minutes), at baseline testing and upon completion of each arm (Days 1, 8, 15).

SECONDARY OUTCOMES:
Diurnal and prandial variation of GLP-1 will correlate with improved glycemia (serum glucose measured in mg/dL) in the eTRE arm | Day 1 through Day 15
  Measure of change in diurnal and prandial variation of GLP-1 levels during glucose tolerance test in the eTRE arm relative to the UPF arm between Days1, 8, and 15.
Diurnal and fasting variation of beta-hydroxybutyrate will correlate with improved glycemia (glucose levels measured in mg/dL) in the eTRE arm | Day 1 through Day 15
  Measure of change fasting beta-hydroxybutyrate levels in the eTRE arm relative to the UPF arm between Days 1, 8, and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Aleman, MD, PhD, Principal Investigator — The Rockefeller University Hospital
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article after deidentification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning one year after publication, no end date
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be sent to jaleman@rockefeller.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Background] Bruno J, Walker JM, Nasserifar S, Upadhyay D, Ronning A, Vanegas SM, Popp CJ, Barua S, Aleman JO. Weight-neutral early time-restricted eating improves glycemic variation and time in range without changes in inflammatory markers. iScience. 2024 Nov 29;27(12):111501. doi: 10.1016/j.isci.2024.111501. eCollection 2024 Dec 20. PMID 39759025
- [Background] Aleman JO, Iyengar NM, Walker JM, Milne GL, Da Rosa JC, Liang Y, Giri DD, Zhou XK, Pollak MN, Hudis CA, Breslow JL, Holt PR, Dannenberg AJ. Effects of Rapid Weight Loss on Systemic and Adipose Tissue Inflammation and Metabolism in Obese Postmenopausal Women. J Endocr Soc. 2017 Apr 25;1(6):625-637. doi: 10.1210/js.2017-00020. eCollection 2017 Jun 1. PMID 29264516
- [Background] Bruno J, Verano M, Vanegas SM, Weinshel E, Ren-Fielding C, Lofton H, Fielding G, Schwack B, Chua DL, Wang C, Li H, Aleman JO. Body Weight and Prandial Variation of Plasma Metabolites in Subjects Undergoing Gastric Band-Induced Weight Loss. Obes Med. 2022 Aug;33:100434. doi: 10.1016/j.obmed.2022.100434. Epub 2022 Jul 1. PMID 37216066
- [Background] Wilkinson MJ, Manoogian ENC, Zadourian A, Lo H, Fakhouri S, Shoghi A, Wang X, Fleischer JG, Navlakha S, Panda S, Taub PR. Ten-Hour Time-Restricted Eating Reduces Weight, Blood Pressure, and Atherogenic Lipids in Patients with Metabolic Syndrome. Cell Metab. 2020 Jan 7;31(1):92-104.e5. doi: 10.1016/j.cmet.2019.11.004. Epub 2019 Dec 5. PMID 31813824
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Scheer FA, Hilton MF, Mantzoros CS, Shea SA. Adverse metabolic and cardiovascular consequences of circadian misalignment. Proc Natl Acad Sci U S A. 2009 Mar 17;106(11):4453-8. doi: 10.1073/pnas.0808180106. Epub 2009 Mar 2. PMID 19255424
- [Background] Sakai R, Hashimoto Y, Ushigome E, Miki A, Okamura T, Matsugasumi M, Fukuda T, Majima S, Matsumoto S, Senmaru T, Hamaguchi M, Tanaka M, Asano M, Yamazaki M, Oda Y, Fukui M. Late-night-dinner is associated with poor glycemic control in people with type 2 diabetes: The KAMOGAWA-DM cohort study. Endocr J. 2018 Apr 26;65(4):395-402. doi: 10.1507/endocrj.EJ17-0414. Epub 2018 Jan 27. PMID 29375081
- [Background] Poggiogalle E, Jamshed H, Peterson CM. Circadian regulation of glucose, lipid, and energy metabolism in humans. Metabolism. 2018 Jul;84:11-27. doi: 10.1016/j.metabol.2017.11.017. Epub 2018 Jan 9. PMID 29195759
- [Background] Morris CJ, Yang JN, Garcia JI, Myers S, Bozzi I, Wang W, Buxton OM, Shea SA, Scheer FA. Endogenous circadian system and circadian misalignment impact glucose tolerance via separate mechanisms in humans. Proc Natl Acad Sci U S A. 2015 Apr 28;112(17):E2225-34. doi: 10.1073/pnas.1418955112. Epub 2015 Apr 13. PMID 25870289
- [Background] McHill AW, Phillips AJ, Czeisler CA, Keating L, Yee K, Barger LK, Garaulet M, Scheer FA, Klerman EB. Later circadian timing of food intake is associated with increased body fat. Am J Clin Nutr. 2017 Nov;106(5):1213-1219. doi: 10.3945/ajcn.117.161588. Epub 2017 Sep 6. PMID 28877894
- [Background] Jones R, Pabla P, Mallinson J, Nixon A, Taylor T, Bennett A, Tsintzas K. Two weeks of early time-restricted feeding (eTRF) improves skeletal muscle insulin and anabolic sensitivity in healthy men. Am J Clin Nutr. 2020 Oct 1;112(4):1015-1028. doi: 10.1093/ajcn/nqaa192. PMID 32729615
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- See also: Research on the positive effect of Time Restricted Feeding (TRF) on hyperglycemia and glucose control. — https://www.healthline.com